CLINICAL TRIAL: NCT02199197
Title: A Phase 2 Randomized Study Comparing Radium Ra 223 Dichloride Plus Enzalutamide With Enzalutamide Alone in Men With Metastatic Castration Refractory Prostate Cancer
Brief Title: Radium Ra 223 With Enzalutamide Compared to Enzalutamide Alone in Men With Metastatic Castration Refractory Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCI68770
Record Dates: First submitted 2014-04-22; First posted 2014-07-24 (Estimated); Results first posted 2019-05-21 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — radium Ra 223 dichloride; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radium Ra 223 Dichloride and Enzalutamide (Experimental): Radium Ra 223 Dichloride and Enzalutamide administered concurrently for 6 28-day cycles.
  Interventions: Drug: Radium Ra 223 Dichloride; Drug: Enzalutamide
- Enzalutamide alone (Active Comparator): Enzalutamide administered as a single agent for 6 28-day cycles.
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Radium Ra 223 Dichloride — Radium Ra 223 Dichloride, 55 kilobecquerel (kBq)/kg body weight, administered as a bolus intravenous (IV) injection (up to 1 minute) on Day 1 of each cycle for 6 cycles.
  Other Names: Xofigo; Alpharadin
  Arms: Radium Ra 223 Dichloride and Enzalutamide
Drug: Enzalutamide — Enzalutamide 160 mg administered orally once a day (continuously) for 6 cycles.
  Other Names: Xtandi

SUMMARY:
Study of Radium Ra 223 dichloride with enzalutamide compared to enzalutamide alone in men with metastatic castration refractory prostate cancer

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented adenocarcinoma of the prostate.
* Men at least 18 years of age and life expectancy of greater than or equal to 6 months.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.
* Metastatic disease as evidenced by both lymphadenopathy and bony metastases or just bony metastases on baseline bone scan and/or computed tomography (CT) scan or MRI of the abdomen and pelvis within 28 days of registration. Chest imaging is only required if clinically indicated or if there is known disease in the chest.
* Castration resistant prostatic adenocarcinoma. Subjects must have castrate levels of serum testosterone (less than 50 ng/dL) achieved by orchiectomy or luteinizing hormone-releasing hormone (LHRH) agonist or antagonist therapy.
* Previously received docetaxel or are not healthy enough per clinical judgment or declined to receive it
* Evidence of disease progression on or after the most recent systemic treatment defined by the following criteria:

  * Prostate-Specific Antigen (PSA): Increasing serum PSA levels as defined by the Prostate Cancer Working Group 2 (PCWG2), determined by 2 consecutive measurements (compared to a baseline or nadir value). If the third measurement is below the second, then a fourth measurement must be greater than the second. The confirming third or fourth measurement must be greater or equal to 2 ng/mL. PSA progression must have occurred within 15 months of registration (with at least 7 days between each PSA measurement). Additionally, the PSA progression as described above should have occurred during or after the most recent systemic treatment for prostate cancer.
  * Measurable disease: greater than or equal to 20% increase in the sum of the short axis diameter of all measurable lymph nodes or the development of any new measurable lymphadenopathy by RECIST 1.1 and PCWG2 criteria.
  * Non-measurable disease:
* Lymph node disease: The appearance of 1 or more new lymphadenopathy, and/or unequivocal worsening of non-measurable disease when compared to imaging studies acquired during castration therapy or against the pre-castration studies if there was no response.
* Bone disease: Appearance of 2 or more new areas of abnormal uptake on bone scan when compared to imaging studies acquired during castration therapy or against the pre-castration studies if there was no response. Increased uptake of pre-existing lesions on bone scan does not constitute progression.
* Symptomatic bone metastases
* Adequate hematologic, renal, and liver function as evidenced by laboratory test results. (Transfusion of blood products are not allowed to normalize blood parameters within 4 weeks of the first radium treatment.)
* Subjects who have previously received docetaxel or are ineligible for docetaxel and who are candidates for treatment with enzalutamide alone or enzalutamide in combination with Radium-223
* Men must agree to use adequate contraception beginning at the signing of the Informed Consent Form until at least 6 months after the last dose of study drug. Because of the potential side effect on spermatogenesis associated with radiation, men who are sexually active must agree to use condoms and their female partners of reproductive potential must agree to use a highly effective contraceptive method during and for 6 months after completing treatment.
* Able to provide informed consent and have signed an approved consent form that conforms to federal and institutional guidelines to ensure compliance with HIPAA regulations.

Exclusion Criteria:

* The presence of known brain metastases, malignant pleural effusions, or malignant ascites. Brain MRI is required at screening only if clinically indicated.
* Visceral metastases as assessed by chest, abdominal or pelvic computed tomography (CT) (or other imaging modality)
* Received systemic therapy with radionuclides (e.g., strontium-89, samarium-153, rhenium-186, or rhenium-188, or Radium Ra 223 dichloride) for the treatment of bony metastases
* Prior treatment with enzalutamide.
* Concurrent anti-cancer therapy (chemotherapy, radiation therapy, surgery, immunotherapy, biologic therapy, or tumor embolization) other than the protocol based treatment. LHRH agonist or antagonist therapy, and supportive non-cancer directed therapies like bisphosphonates or denosumab are allowed.
* Prior cytoxic chemotherapy with the exception of docetaxel or cabazitaxel. Treatment with docetaxel or cabazitaxel must be discontinued greater than 4 weeks from the time of enrollment, and recovery of adverse events (AEs) to grade 1 or baseline (however, ongoing neuropathy is permitted).
* Major surgery within 30 days prior to start of study drug
* Current, untreated pathologic long-bone fractures, imminent pathologic long-bone fractures (cortical erosion on radiography greater than 50%).
* Prior hemi-body external radiotherapy. Subjects who received other types of prior external radiotherapy are allowed provided that bone marrow function is assessed and meets the protocol requirements for hemoglobin, absolute neutrophil count (ANC), and platelets.
* Use of biologic response modifiers, such as granulocyte macrophage colony-stimulating factor (GM-CSF) or granulocyte colony-stimulating factor (G-CSF) within 4 weeks prior to screening
* Lymphadenopathy exceeding 3 cm in short-axis diameter
* Any size pelvic lymphadenopathy if it is thought to be a contributor to concurrent hydronephrosis.
* Current or imminent spinal cord compression based on clinical findings and/or magnetic resonance imaging (MRI). Treatment should be completed for spinal cord compression.
* Any other serious illness or medical condition in the opinion of the investigator, such as but not limited to:
* Any greater than or equal to Grade 2 infection as defined by NCI-CTCAE version 4.03.
* Cardiac failure New York Heart Association (NYHA) III or IV
* Crohn's disease or ulcerative colitis
* Bone marrow dysplasia
* Fecal incontinence
* Concomitant use of narrow therapeutic index drugs that are metabolized by CYP3A4 (i.e. alfentanil, cyclosporine, dihydroergotamine, ergotamine, fentanyl, pimozide, quinidine, sirolimus, tacrolimus), CYP2C9 (phenytoin, warfarin), and CYP2C19 (S-mephenytoin). [Note: Patients on stable doses of anti-coagulation with warfarin and fentanyl will be eligible, as long as they are monitored closely with additional international normalized ratio (INR) monitoring].
* Any infection requiring parenteral antibiotic therapy or causing fever (temperature greater than 100.5 degrees F or 38.1 degrees C) within 1 week prior to registration.
* Concurrent other malignancy with the exception of: a) cutaneous squamous cell and basal carcinomas, b) adequately treated stage 1-2 malignancy , c) adequately treated stage 3-4 malignancy that had been in remission for greater than or equal to 2 years at the time of registration.
* Inability to comply with the protocol and/or not willing or not available for follow-up assessments
* Any medical intervention or other condition which, in the opinion of the Principal Investigator could compromise adherence with study requirements or otherwise compromise the study's objectives

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2014-06-25 (Actual); Primary Completion 2018-04-19 (Actual); Study Completion 2019-10-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Agarwal N, Nussenzveig R, Hahn AW, Hoffman JM, Morton K, Gupta S, Batten J, Thorley J, Hawks J, Santos VS, Nachaegari G, Wang X, Boucher K, Haaland B, Maughan BL. Prospective Evaluation of Bone Metabolic Markers as Surrogate Markers of Response to Radium-223 Therapy in Metastatic Castration-resistant Prostate Cancer. Clin Cancer Res. 2020 May 1;26(9):2104-2110. doi: 10.1158/1078-0432.CCR-19-2591. Epub 2020 Jan 14. PMID 31937614

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radium Ra 223 Dichloride and Enzalutamide | Enzalutamide Alone
Started | 35 | 14
Completed | 35 | 12
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Radium Ra 223 Dichloride and Enzalutamide: Radium Ra 223 Dichloride and Enzalutamide administered concurrently for 6 28-day cycles.
  Radium Ra 223 Dichloride: Radium Ra 223 Dichloride, 55 kBq/kg body weight, administered as a bolus intravenous (IV) injection (up to 1 minute) on Day 1 of each cycle for 6 cycles.
  Enzalutamide: Enzalutamide 160 mg administered orally once a day (continuously) for 6 cycles.
- Total: Total of all reporting groups
Arm/Group | Radium Ra 223 Dichloride and Enzalutamide | Enzalutamide Alone | Total
Number analyzed (Participants) | 35 | 14 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 5 | 16
  >=65 years | 24 | 9 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.66 (8.20) | 68.64 (8.04) | 68.65 (8.07)
Age, Continuous [Median (Full Range); unit: years] | 69 [55 to 85] | 69.5 [54 to 81] | 69 [54 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 35 | 14 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 34 | 14 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 34 | 14 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Serum N-Telopeptide Levels (Log2 scale) [Mean (Full Range); unit: nM BCE] — Population: Two patients on the Enzalutamide only arm did not have subsequent N-Telopeptide labs drawn and were excluded from the N-Telopeptide analysis, so are excluded here as well.
  nM BCE
    number analyzed (Participants) | 35 | 12 | 47
    (all) | 3.42 [2.41 to 4.68] | 3.41 [2.77 to 4.3] | 3.42 [2.41 to 4.68]

OUTCOME MEASURES:

1. Primary Outcome: Fold Change in Serum N-telopeptides From Baseline
Description: Patients had serum N-telopeptide labs drawn prior to the start of treatment and at the End of Treatment visit or at disease progression, whichever occurred first. The mean and standard deviation of the differences were calculated on a log 2 scale. Fold changes (post/pre) and 95% confidence intervals are reported.
Time Frame: From prior to start of treatment to end of treatment or disease progression (approximately 6 months)
Population: Per study protocol, only randomized patients with bone marker level measurements at baseline and Cycle 3 Day 1 will be evaluable for the primary efficacy outcome. 8 patients were assigned to Radium + Enzalutamide without randomization and were excluded from analysis. 2 patients on Enzalutamide alone did not reach Cycle 3 Day 1 and were excluded.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Radium Ra 223 Dichloride and Enzalutamide | Enzalutamide Alone
Number analyzed (Participants) | 27 | 12
fold change | 0.85 [0.76 to 0.94] | 1.34 [0.99 to 1.81]

2. Primary Outcome: Number of Participants With Adverse Events
Description: Adverse Events were assessed from start of Radium Ra 223 Dichloride or Enzalutamide treatment (whichever was started first) through 30 days after the last dose of either drug or until start of a new anti-cancer therapy, whichever came first. Adverse events were assessed using the Common Terminology for Adverse Events (CTCAE) version 4.0. Each event was assigned a grade (1-5), with lower grades indicating milder events. All adverse events were recorded, regardless of attribution to study treatment. Reported below are the number of patients who experienced any grade 3-5 non-hematological AE. A full listing of AEs affecting 5% or more participants are listed in the Adverse Events module of the Results section.
Time Frame: From first dose of study treatment to 30 days following last dose (approximately 7 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Radium Ra 223 Dichloride and Enzalutamide | Enzalutamide Alone
Number analyzed (Participants) | 35 | 14
Participants | 9 | 2

3. Secondary Outcome: Prostate Specific Antigen (PSA) Progression Free Survival (PFS)
Description: Prostate Specific Antigen (PSA) Progression Free Survival (PFS) is the time during with participants did not experience PSA progression. This is measured from the start of study therapy to the time of PSA progression. PSA progression is defined as a rise in PSA of at least 25% and at least 2 ng/ml from baseline or nadir. Kaplan-Meier methods were used.
Time Frame: Up to 2 years (24 months)
Population: Two participants who dropped out prior to Cycle 3 were excluded from analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Radium Ra 223 Dichloride and Enzalutamide | Enzalutamide Alone
Number analyzed (Participants) | 35 | 12
months | 9.86 [4.67 to 22.5] | 3.34 [2.66 to NA] — Value is infinity because there were too few participants to get a real number.

4. Secondary Outcome: Radiographic Progression Free Survival (PFS)
Description: Radiographic Progression Free Survival (PFS) is the time during with participants did not experience disease progression based on study imaging. This is measured from the start of study therapy to the time of radiographic progression. Radiographic progression was defined by the Prostate Cancer Working Group 2 (PCWG2) criteria, in which soft tissue disease is evaluated by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and bone lesions are evaluated separately under PCWG2 criteria. PCWG2 and RECIST 1.1 are established radiographic assessment protocols. Kaplan-Meier methods were used.
Time Frame: Up to 2 years (24 months)
Population: Two participants who dropped out prior to Cycle 3 were excluded from analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Radium Ra 223 Dichloride and Enzalutamide | Enzalutamide Alone
Number analyzed (Participants) | 35 | 12
months | 11.31 [9.07 to NA] — Value is infinity because there were too few participants to get a real number. | 5.62 [2.76 to NA] — Value is infinity because there were too few participants to get a real number.

5. Secondary Outcome: Bone Alkaline Phosphatase (ALP) Progression Free Survival (PFS)
Description: Bone Alkaline Phosphatase (ALP) Progression Free Survival (PFS) is the time during with participants did not experience Bone ALP progression. This is measured from the start of study therapy to the time of Bone ALP progression. Bone ALP progression defined as a rise in Bone ALP of at least 25% and at least 2 micrograms (mcg)/L from baseline or nadir. Kaplan-Meier methods were used.
Time Frame: Up to 2 years (24 months)
Population: Two participants who dropped out prior to Cycle 3 were excluded from analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Radium Ra 223 Dichloride and Enzalutamide | Enzalutamide Alone
Number analyzed (Participants) | 35 | 12
months | NA [NA to NA] — Too few participants demonstrated Bone ALP progression to obtain a median, and thus 95% confidence intervals are infinite. | 4.64 [2.76 to NA] — Value is infinity because there were too few participants to get a real number.

6. Secondary Outcome: Count of Prostate Specific Antigen (PSA) Responses
Description: Prostate Specific Antigen (PSA) Responses in participants were categorized based on decrease from baseline: less than 30% (<30%) decrease (including increases from baseline), greater than or equal to 30% (>=30%) decrease, greater than or equal to 50% (>=50%) decrease, and greater than or equal to 90% (>=90%) decrease. Count of participants in each category are provided
Time Frame: Up to 2 years after start of study treatment
Population: Two participants who dropped out prior to Cycle 3 were excluded from analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Radium Ra 223 Dichloride and Enzalutamide | Enzalutamide Alone
Number analyzed (Participants) | 35 | 12
Participants
  <30% | 6 | 6
  >=30% | 5 | 2
  >=50% | 9 | 2
  >=90% | 15 | 2

7. Secondary Outcome: Count of Radiographic Responses
Description: Radiographic Responses in participants were assessed using the Prostate Cancer Working Group 2 (PCWG2) criteria. Possible responses include Complete Response (CR) (complete disappearance of all metastatic disease on imaging), Partial Response (PR) (improvement in metastatic disease on imaging), Stable Disease (SD) (neither worsening nor improvement of metastatic disease on imaging), and Progressive Disease (PD) (worsening of metastatic disease on imaging). A count of participants in each category is provided here.
Time Frame: Up to 2 years after start of study treatment
Population: Two participants who dropped out prior to Cycle 3 were excluded from analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Radium Ra 223 Dichloride and Enzalutamide | Enzalutamide Alone
Number analyzed (Participants) | 35 | 12
Participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 3 | 0
  Stable Disease (SD) | 28 | 8
  Progressive Disease (PD) | 4 | 4

8. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) is the time during which participants did not pass away. This is measured from the start of study therapy to the time of death from any cause. Kaplan-Meier methods were used.
Time Frame: Up to 40 months
Population: Two participants who dropped out prior to Cycle 3 were excluded from analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Radium Ra 223 Dichloride and Enzalutamide | Enzalutamide Alone
Number analyzed (Participants) | 35 | 12
months | 26.0 [17.6 to NA] — Value is infinity because there were too few participants to get a real number. | 21.0 [16.6 to NA] — Value is infinity because there were too few participants to get a real number.

ADVERSE EVENTS:
Time Frame: The collection of adverse events began after the first dose of study treatment and end 30 days after the last dose of study treatment (or until new cancer treatment was initiated, if sooner) (approximately 7 months).
Description: The occurrence of adverse events was sought by non-directive questioning of the patient at each visit or phone contact during the study. Adverse events also may have been detected when they were volunteered by the patient during or between visits or through physical examination, laboratory test, or other assessments.
Arm/Group | Radium Ra 223 Dichloride and Enzalutamide | Enzalutamide Alone
All-Cause Mortality (participants affected / at risk) | 15/35 | 8/14
Serious Adverse Events (participants affected / at risk) | 7/35 | 2/14
Other Adverse Events (participants affected / at risk) | 35/35 | 12/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radium Ra 223 Dichloride and Enzalutamide (N=35) | Enzalutamide Alone (N=14)
Anaphylaxis (Immune system disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 0 — inguinal hernia
Lung infection (Infections and infestations) | 1 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — disease progression - metastatic prostate cancer
Neutrophil count decreased (Investigations) | 1 | 0
Pain (General disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radium Ra 223 Dichloride and Enzalutamide (N=35) | Enzalutamide Alone (N=14)
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Alkaline phosphatase increased (Investigations) | 1 | 3 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 9 (13) | 1
Anorexia (Metabolism and nutrition disorders) | 12 | 0
Anxiety (Psychiatric disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (12) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (9) | 1
Bloating (Gastrointestinal disorders) | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 2
Chills (General disorders) | 2 (3) | 1
Constipation (Gastrointestinal disorders) | 10 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Creatinine increased (Investigations) | 1 (2) | 1 (2)
Depression (Psychiatric disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 19 (25) | 1
Dizziness (Nervous system disorders) | 4 (5) | 0
Dysgeusia (Nervous system disorders) | 5 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 2 | 0 — inner ear "fullness"; "rattling in ears" attributed to hearing loss
Edema limbs (General disorders) | 6 (7) | 0
Facial pain (General disorders) | 0 | 1
Fatigue (General disorders) | 16 (20) | 3
Flatulence (Gastrointestinal disorders) | 1 | 1
Flu like symptoms (General disorders) | 6 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 | 1 — viral syndrome / food poisoning
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 1
Gum infection (Infections and infestations) | 2 | 0
Gynecomastia (Reproductive system and breast disorders) | 0 | 1
Headache (Nervous system disorders) | 5 (6) | 0
Hot flashes (Vascular disorders) | 4 (5) | 0
Hypertension (Vascular disorders) | 3 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 4 | 0
Insomnia (Psychiatric disorders) | 2 | 0
Lymphocyte count decreased (Investigations) | 18 (38) | 4 (6)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 3 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 16 (23) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 — polyps found on colonoscopy; esophageal carcinoma
Neutrophil count decreased (Investigations) | 14 (36) | 0
Non-cardiac chest pain (General disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (8) | 1
Palpitations (Cardiac disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 4 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1
Platelet count decreased (Investigations) | 7 (9) | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 0
Psychiatric disorders - Other (Psychiatric disorders) | 0 | 1 — fuzzy/foggy-headed
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 | 0 — dog bite; hives
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (2)
Syncope (Nervous system disorders) | 2 | 0
Testicular pain (Reproductive system and breast disorders) | 2 | 0
Urinary frequency (Renal and urinary disorders) | 2 | 1
Urinary urgency (Renal and urinary disorders) | 2 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 4 | 0
Weight loss (Investigations) | 4 | 0
White blood cell decreased (Investigations) | 20 (47) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-06): https://cdn.clinicaltrials.gov/large-docs/97/NCT02199197/Prot_SAP_000.pdf